CLINICAL TRIAL: NCT05447481
Title: A Randomized Double-blind, Placebo-controlled, Cross-over Study to Evaluate the Effects of Chicory Inulin-type Fructans in Adults With Functional Constipation
Brief Title: Evaluation of the Effect of Chicory Inulin-type Fructans in Constipated Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensus (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry); Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AFCRO-058
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Constipation - Functional
Keywords: adults; functional constipation; inulin-type fructans

STUDY DESIGN:
Intervention Model Description: This was a randomized, double-blind, placebo-controlled, cross-over study to evaluate the effects of chicory inulin-type fructans in adults with functional constipation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects were blinded to the study treatment that they received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chicory inulin-type fructan - placebo (Experimental): Dietary supplement: chicory inulin-type fructan Placebo: maltodextrin
  Interventions: Dietary Supplement: chicory inulin-type fructan
- Placebo - chicory inulin-type fructan (Experimental): Placebo: maltodextrin Dietary Supplement: chicory inulin-type fructan
  Interventions: Dietary Supplement: chicory inulin-type fructan

INTERVENTIONS:
Dietary Supplement: chicory inulin-type fructan — Dietary supplement: chicory inulin-type fructan

SUMMARY:
Constipation is common in the general population, especially in women and in the elderly, which can significantly affect quality of life of the individual. There is a general consumer trend to seek natural food options, also when addressing health issues such as constipation. Consumers seek tasty options and there is a paucity of tasty functional foods to address constipation. Adding natural fiber to food, like inulin-type fructans from chicory root fiber, can increase fiber intake and potentially prevent or resolve constipation issues. This study aimed to increase the body of scientific data on inulin-type fructans by way of a randomized, placebo-controlled, cross-over study. Maltodextrin was used as the placebo in this study.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent
* Between 18 and 75 years of age
* Have functional constipation according to the Rome III Diagnostic Criteria
* Subjects were to continue on their normal diet and agreed to not take probiotic or prebiotic products/supplements and supplemental dietary fibres for the duration of the study
* The subject agrees to complete the Patient Diary for two weeks prior to study entry and for the duration of the study
* Subject is in general good health as determined by the investigator.

Exclusion Criteria:

* Subjects less than 18 and greater than 75 years of age
* Females who are pregnant, lactating or wish to become pregnant during the study.
* Subjects who are hypersensitive to any of the components of the test product,
* Subjects who have an obstructive or metabolic aetiology for constipation,
* Subjects who have a history of laxative abuse (greater than the daily dosage recommended on the label for any laxative),
* Subjects currently taking supplemental dietary fibres or have taken them within two weeks of the screening visit,
* Subjects who are taking a probiotic or prebiotic product/supplement or had taken them within two weeks of the screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Change in stool frequency | During the 12 week intervention period
  Determine the impact of chicory inulin-type fructan on stool frequency in constipated subjects.

SECONDARY OUTCOMES:
Change in stool consistency | During the 12 week intervention period
  Determine the effect of chicory inulin-type fructans on stool consistency in constipated subjects.
Patient Assessment of Constipation Symptoms | During the 12 week intervention period
  Determine the effect of chicory inulin-type fructans on constipation symptoms using the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire.
Quality of life using the PAC-QOL questionnaire | During the 12 week intervention period
  Determine the effect of chicory inulin-type fructans on quality of life using the PAC-QOL questionnaire
Physical activity | During the 12 week intervention period
  Determine the physical activity of the subjects using the International Physical Activity Questionnaire (IPAQ)
Resort to laxatives | During the 12 week intervention period
  Determine the resort to laxatives of the subjects
Gut microbiota composition | During the 12 week intervention period
  Determine the effect of chicory inulin-type fructans on gut microbiota composition

CONTACTS AND LOCATIONS:
Overall Officials: Elaine E Vaughan, PhD, Study Chair — Sensus BV

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puhlmann ML, Wegh CAM, van der Zalm SCC, Dam V, Doolan A, Meyer D, Belzer C, Vaughan EE, Benninga MA, Smidt H. Inulin-induced improvements on bowel habit and gut microbiota in adults with functional constipation: findings of a randomized, double-blind, placebo-controlled study. BMC Gastroenterol. 2025 Nov 13;25(1):806. doi: 10.1186/s12876-025-04409-6. PMID 41233756